CLINICAL TRIAL: NCT03999060
Title: Brainstem Mapping of Nociceptive Trigeminal Input
Brief Title: Trigeminal Brainstem Mapping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: TrigeminalBrainstemMapping
Record Dates: First submitted 2019-06-13; First posted 2019-06-26 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Headache Disorders, Primary; Migraine
MeSH Terms: conditions — Headache Disorders, Primary; Migraine Disorders | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electric Stimulation (Experimental)
  Interventions: Device: Electric Current Stimulation

INTERVENTIONS:
Device: Electric Current Stimulation — Electric stimulation with a Digitimer DS7AH HV Current Stimulator delivered with 4 shielded electrodes mounted on the participants head

SUMMARY:
To what extent the somatotopy of the 3 branches of the trigeminal nerve (V1,V2,V3) as well as the greater occipital nerve (GON) in the brainstem but also in the thalamus and the insula can be mapped using functional imaging and BOLD in humans is not known but might play an important role in imaging headache diseases. The aim is to map their somatotopy by random stimulation of V1, V2, V3 and the GON with painful electrical input during acquisition of BOLD-fMRI.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* suitable fo MRI

Exclusion Criteria:

* headache disease
* psychological disorder
* pregnancy
* all exclusion criteria necessary for imaging in a 3 T MRI scanner

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-06-28 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Statistical Parametric Map calculated from the fMRI data on brainstem level | through study completion, an average of 9 months
  At a statistical threshold of T-value 3 we will observe a somatotopical arrangement in the brainstem below the pons:
  Expected location for V1: within radius of 10 mm around the MNI coordinates (-1,-48,-75); Expected location for V2: within radius of 10 mm around the MNI coordinates (-4,-47,-69) Expected location for V3: within radius of 10 mm around the MNI coordinates (-1,-46,-66) Expected location for GON: within radius of 10 mm around the MNI coordinates (-1,-45,-64)
Statistical Parametric Map calculated from the fMRI data in the thalamus | through study completion, an average of 9 months
  At a statistical threshold of T-value 4 we will observe a somatotopical arrangement in the thalamus:
  Expected location for V1: within radius of 10 mm around the MNI coordinates (11,-5,6); Expected location for V2: within radius of 10 mm around the MNI coordinates (13,-11,5) Expected location for V3: within radius of 10 mm around the MNI coordinates (12,-10,5) Expected location for GON: within radius of 10 mm around the MNI coordinates (15,-12,-7)
Statistical Parametric Map calculated from the fMRI data in the insula | through study completion, an average of 9 months
  At a statistical threshold of T-value 4 we will observe a somatotopical arrangement in the insula:
  Expected location for V1: within radius of 10 mm around the MNI coordinates (38,-15,8); Expected location for V2: within radius of 10 mm around the MNI coordinates (37,-8,-5) Expected location for V3: within radius of 10 mm around the MNI coordinates (39,2,-11) Expected location for GON: within radius of 10 mm around the MNI coordinates (38,-12,-3)

SECONDARY OUTCOMES:
Statistical Parametric Map calculated from the fMRI data in the cerebellum | through study completion, an average of 9 months
Statistical Parametric Map calculated from the fMRI data in the periaqueductal gray (PAG) | through study completion, an average of 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Arne May, Prof. Dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- UKE, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No
Group results will be presented at international conferences as well as published in international peer-reviewed journals

REFERENCES:
- [Derived] Mehnert J, Basedau H, Sturm LM, Nielsen T, Jensen RH, May A. Functional brainstem representations of the human trigeminal cervical complex. Cephalalgia. 2023 May;43(5):3331024231174862. doi: 10.1177/03331024231174862. PMID 37203351